CLINICAL TRIAL: NCT00999024
Title: Reflectometric Measurement of Retinal Oxygen Saturation in Patients With COPD Grade IV and Healthy Subjects
Brief Title: Reflectometric Measurement of Retinal Oxygen Saturation in Patients With Chronic Obstructive Pulmonary Disease (COPD) Grade IV and Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gerhard Garhofer, MD, Department of Clinical Pharmacology, Medical University of Vienna
Other Study IDs: OPHT - 090709
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2009-10

CONDITIONS: Retinal Artery; Retinal Veins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy subjects: 20 healthy subjects will be included
- COPD Patients: 20 Patients with Grade IV COPD will be included

SUMMARY:
An adequate oxygenation and retinal perfusion is essential for the function of the inner retina. There is a wide range of autoregulation mechanisms to ensure a sufficient ocular blood and oxygen supply during changes in systemic blood pressure or intraocular pressure (IOP). Nonetheless, various retinopathies such as diabetic retinopathy, which is the leading cause of blindness in people aged 20-65 in the western world, are highly associated with hypoxia (Pemp and Schmetterer 2008). Hence, measurements of oxygen levels in retinal vessels are needed to further our understanding of these ischemic diseases. It is a well known fact and a commonly employed method to measure oxygen saturation of blood through light transmission (Kramer 1934). However, this approach is not feasible in the human eye. Therefore, reflection must be used, meaning the amount of incident light must be estimated based on the amount of light reflected (for a review see Harris 2003). This is a difficult task and investigators in this field have encountered several problems, including optical complexities, nonlinear sensors and eye movement (Beach et al 1999; Delori 1988). Nonetheless considerable progress has been made over the past decades and the development of an reliable oximeter reported (Hardarson et al 2006).

In the present study this technique will be applied in healthy subjects as well as in patients with COPD during room-air conditions. The procedure takes approximately 15 minutes in each subject and will be performed in only one eye.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for healthy subjects:

* Men and women aged between 18 and 99 years
* Tiffeneau Index > 70 %
* Body mass index between 15th and 85th percentile
* Normal ophthalmic findings, ametropia < 3 Dpt.

Inclusion criteria for COPD patients:

* Men and women aged between 18 and 99 years
* COPD grade IV, oxygen dependent and with a forced expiratory volume in 1 second (FEV1) < 30 %
* Body mass index between 15th and 85th percentile
* Normal ophthalmic findings, ametropia < 3 Dpt.

Exclusion Criteria:

Healthy subjects:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug except oral contraceptives
* Symptoms of a clinically relevant illness in the 3 weeks before the study day
* Blood donation during the previous 3 weeks

COPD patients:

* Abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Health status which does interfere with study procedure or their safety
* Blood donation during the previous 3 weeks
* Symptoms of a clinically relevant illness other than COPD or COPD related in the 3 weeks before the study day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 healthy subjects, 20 patients with grade IV COPD
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Blood oxygen saturation measured in retinal vessel | 15 minutes measured with the RVA

SECONDARY OUTCOMES:
Systemic blood pressure | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhofer, MD, Priv.Doz., Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Palkovits S, Lasta M, Boltz A, Schmidl D, Kaya S, Hammer M, Marzluf B, Popa-Cherecheanu A, Frantal S, Schmetterer L, Garhofer G. Measurement of retinal oxygen saturation in patients with chronic obstructive pulmonary disease. Invest Ophthalmol Vis Sci. 2013 Feb 5;54(2):1008-13. doi: 10.1167/iovs.12-10504. PMID 23307953